CLINICAL TRIAL: NCT03189173
Title: Combined Upper-airway and Breathing Control Therapies for Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Monash University (Other); American Heart Association (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Heart Foundation of Australia (Unknown)
Responsible Party: Principal Investigator, Scott Aaron Sands, Associate Physiologist / Instructor in Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P001037; 15SDG25890059 (Other Grant/Funding Number: American Heart Association); R01HL128658 (NIH)
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Ventilatory Control Instability; Complex Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Occlusal Splints; Oxygen; Combined Modality Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Subjects will receive mandibular advancement, supplemental oxygen, mandibular advancement plus supplemental oxygen, and no treatment in randomized order. On nights without supplemental oxygen, subjects will be administered sham (air, single blinded). Oral appliance use will not be masked.
Who Masked: Participant, Outcomes Assessor
Masking Description: Supplemental oxygen versus air assignment nights will be blinded to participants, but will be known by the investigator. Oral appliances will be "open label".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (20):
- Combo, Mad, Sham, Oxygen (Experimental): Order of interventions: Combo, Mad, Sham, Oxygen
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Combo, Oxygen, Mad, Sham (Experimental): Order of interventions: Combo, Oxygen, Mad, Sham
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Combo, Oxygen, Sham, MAD (Experimental): Order of interventions: Combo, Oxygen, Sham, MAD
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Combo, Sham, Mad, Oxygen (Experimental): Order of interventions: Combo, Sham, Mad, Oxygen
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Combo, Sham, Oxygen, MAD (Experimental): Order of interventions: Combo, Sham, Oxygen, MAD
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- MAD, Combo, Oxygen, Sham (Experimental): Order of interventions: MAD, Combo, Oxygen, Sham
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- MAD, Combo, Sham, Oxygen (Experimental): Order of interventions: MAD, Combo, Sham, Oxygen
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- MAD, Oxygen, Combo, Sham (Experimental): Order of interventions: MAD, Oxygen, Combo, Sham
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- MAD, Oxygen, Sham, Combo (Experimental): Order of interventions: MAD, Oxygen, Sham, Combo
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- MAD, Sham, Combo, Oxygen (Experimental): Order of interventions: MAD, Sham, Combo, Oxygen
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- MAD, Sham, Oxygen, Combo (Experimental): Order of interventions: MAD, Sham, Oxygen, Combo
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Oxygen, Combo, Sham, MAD (Experimental): Order of interventions: Oxygen, Combo, Sham, MAD
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Oxygen, MAD, Sham, Combo (Experimental): Order of interventions: Oxygen, MAD, Sham, Combo
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Oxygen, Sham, Combo, MAD (Experimental): Order of interventions: Oxygen, Sham, Combo, MAD
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Oxygen, Sham, MAD, Combo (Experimental): Order of interventions: Oxygen, Sham, MAD, Combo
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Sham, Combo, MAD, Oxygen (Experimental): Order of interventions: Sham, Combo, MAD, Oxygen
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Sham, MAD, Combo, Oxygen (Experimental): Order of interventions: Sham, MAD, Combo, Oxygen
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Sham, MAD, Oxygen, Combo (Experimental): Order of interventions: Sham, MAD, Oxygen, Combo
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Sham, Oxygen, Combo, MAD (Experimental): Order of interventions: Sham, Oxygen, Combo, MAD
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment
- Sham, Oxygen, MAD, Combo (Experimental): Order of interventions: Sham, Oxygen, MAD, Combo
  Interventions: Device: Oral appliance; Drug: Oxygen; Other: Oral appliance plus oxygen; Other: No treatment

INTERVENTIONS:
Device: Oral appliance — An oral appliance (dental mouthpiece) will be used to improve upper airway patency. Patients who do not have their own custom dental oral appliance (various brands, commonly Herbst/Somnomed) will be provided with a device (BluePro, BlueSom) for the duration of the study.
  Patients will also be administered sham (room air) at 4 L/min via nasal cannula.
  Other Names: Mandibular advancement device
Drug: Oxygen — Supplemental oxygen will be delivered at 4 L/min via nasal cannula to improve ventilatory control stability.
  Other Names: Supplemental inspired oxygen
Other: Oral appliance plus oxygen — Both treatments will be administered simultaneously.
  Other Names: Combination therapy
Other: No treatment — Subjects will not wear an oral appliance, and will be administered sham (room air) at 4 L/min via nasal cannula.
  Other Names: Sham

SUMMARY:
The current study combines two treatments for obstructive sleep apnea (OSA), oral appliances and supplemental inspired oxygen. The following aims will be tested:

Aim 1. To determine whether supplemental inspired oxygen further reduces OSA severity (apnea-hypopnea index) in patients using an oral appliance.

Aim 2. To determine whether baseline OSA phenotypes can predict the efficacy of oral appliances versus supplemental oxygen versus both treatments in combination. We will test whether responders to oral appliances have distinct pathophysiological characteristics compared with oxygen responders.

DETAILED DESCRIPTION:
Pre-specified primary analysis for Aim 1 is the change in AHI with combination treatment versus oral appliance alone (%reduction versus placebo; including hypopnea events without desaturation/arousals).

Aim 2 seeks to identify subgroups of patients that have the greatest reduction in AHI (responders) with each treatment (post-hoc). We will use baseline physiological measures of the four traits causing OSA (collapsibility, responsiveness, loop gain, arousal threshold) to determine which characteristics predict responses to each intervention (leave-one-out support vector machine modeling). Clinical measures of the same traits will be estimated from the placebo night to confirm that responses can be predicted with clinically-available data. We will also test whether responders to oral appliances have a greater response to oxygen than oral appliance non-responders (and vice-versa), to address whether responders to both treatments are similar or different.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed OSA or suspected OSA based on snoring

Exclusion Criteria:

* Severe co-morbidities (cardiovascular, renal, lung disease, neurological), including:

Congestive heart failure, Neurological conditions that may affect sleep or breathing (e.g. neuromuscular diseases e.g. myasthenia gravis; neurodegenerative diseases e.g. Alzheimer's/Parkinson's)

* Medications that will substantially affect respiration, including opioids, barbiturates, theophylline, doxapram, acetazolamide, pseudoephedrine
* Claustrophobia
* Insomnia and other non-respiratory sleep disorders
* Inability to sleep supine
* Contraindications to oral appliances, including insufficient teeth to support the device, periodontal problems inducing tooth mobility, active temporomandibular joint disorder
* Allergy to lidocaine or oxymetazoline HCl

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in apnea hypopnea index (AHI), percent of baseline. | Single night
  Primary test is difference between combination therapy and oral appliance

SECONDARY OUTCOMES:
Change in frequency of arousals, percent of baseline. | Single night
  Primary test is difference between combination therapy and oral appliance
Patient reported sleep quality (visual analog scale) | Single night
  Primary test is difference between combination therapy and oral appliance
Morning minus evening systolic blood pressure | Single night
  Primary test is difference between combination therapy and oral appliance
Morning minus evening diastolic blood pressure | Single night
  Primary test is difference between combination therapy and oral appliance

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sands, PhD, Principal Investigator — Brigham and Women's Hospital; Bradley A Edwards, PhD, Principal Investigator — Monash University
Locations (2):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- Sleep and Circadian Medicine Laboratory, BASE Facility, Monash University, Notting Hill, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified subject data will be shared via an online repository.
Time Frame: 6 months after publication

REFERENCES:
- [Derived] Hynes DJ, Mann DL, Landry SA, Joosten SA, Edwards BA, Hamilton GS. Night-to-night variability in obstructive sleep apnea severity, the physiological endotypes, and the frequency of flow limitation. Sleep. 2025 Apr 11;48(4):zsae295. doi: 10.1093/sleep/zsae295. PMID 39688178